CLINICAL TRIAL: NCT01712490
Title: A Randomized, Open-label, Phase 3 Trial of A+AVD Versus ABVD as Frontline Therapy in Patients With Advanced Classical Hodgkin Lymphoma
Brief Title: A Frontline Therapy Trial in Participants With Advanced Classical Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C25003; 2011-005450-60 (EudraCT Number); U1111-1161-4937 (Registry Identifier: WHO); 12/LO/1950 (Registry Identifier: NRES); JapicCTI-142491 (Registry Identifier: JapicCTI); REec-2013-0114 (Registry Identifier: REec); 1025002760 (Registry Identifier: TCTIN); C25003CTID (Other: Israel); 2023-506419-16-00 (EU CTIS Number: EU CTIS)
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Results first posted 2018-11-27 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma; Hodgkins Lymphoma; Antibody, Monoclonal; Antibody-Drug Conjugate; Antigens, CD-30; Immunotherapy; Lymphoma; Lymphoma, Classical; ECHELON-1
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — Brentuximab Vedotin; Doxorubicin; Bleomycin; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A + AVD (Experimental): A+AVD consists of brentuximab vedotin (ADCETRIS®) 1.2 milligram per kilogram (mg/kg) plus doxorubicin 25 milligram per square meter (mg/m^2), vinblastine 6 mg/m^2, and dacarbazine (DTIC) 375 mg/m^2.
  Interventions: Drug: brentuximab vedotin; Drug: doxorubicin; Drug: vinblastine; Drug: dacarbazine
- ABVD (Active Comparator): ABVD consists of doxorubicin 25 mg/m^2, bleomycin 10 units per square meter (units/m^2), vinblastine 6 mg/m^2, and dacarbazine (DTIC) 375 mg/m^2.
  Interventions: Drug: doxorubicin; Drug: bleomycin; Drug: vinblastine; Drug: dacarbazine

INTERVENTIONS:
Drug: brentuximab vedotin — Brentuximab vedotin (ADCETRIS®)1.2 mg/kg by IV infusion on Days 1 and 15 of each 28-day cycle.
  Other Names: ADCETRIS®; SGN-35
  Arms: A + AVD
Drug: doxorubicin — Doxorubicin: 25 mg/m^2 by IV infusion on Days 1 and 15 of each 28-day cycle.
  Other Names: Adriamycin
Drug: bleomycin — Bleomycin: 10 units/m^2 by IV infusion on Days 1 and 15 of each 28-day cycle.
  Arms: ABVD
Drug: vinblastine — Vinblastine: 6 mg/m2 will be administered by IV infusion on Days 1 and 15 of each 28-day cycle
Drug: dacarbazine — Dacarbazine (DTIC): 375 mg/m^2 by IV infusion on Days 1 and 15 of each 28-day cycle.
  Other Names: DTIC

SUMMARY:
This open-label, randomized, 2-arm, multicenter, phase 3 study has the primary objective of comparing the modified progression-free survival (mPFS) obtained with brentuximab vedotin (ADCETRIS®) plus AVD (doxorubicin [Adriamycin], vinblastine, and dacarbazine; abbreviated A+AVD) versus that obtained with ABVD (doxorubicin [Adriamycin],bleomycin, vinblastine, and dacarbazine) for the frontline treatment of advanced classical Hodgkin lymphoma(HL)

ELIGIBILITY:
Inclusion Criteria:

1. Treatment-naïve participants with Ann Arbor Stage III or IV HL.
2. Histologically confirmed classical Hodgkin Lymphoma (HL) according to the current World Health Organization (WHO) classification.
3. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (<=) 2.
4. Bidimensional measurable disease as documented by radiographic technique per the International Working Group Revised Criteria for Response Assessment for Malignant Lymphoma.

Exclusion Criteria:

1. Nodular lymphocyte predominant Hodgkin lymphoma.
2. Cerebral/meningeal disease, including signs and symptoms of progressive multifocalleukoencephalopathy (PML).
3. Sensory or motor peripheral neuropathy.
4. Prior immunosuppressive chemotherapy, therapeutic radiation, or any immunotherapy within 12 weeks of first study drug dose.
5. Known human immunodeficiency virus (HIV) positive.
6. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection.

Please note that there are additional exclusion criteria. The study center will determine if you meet all of the criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1334 (Actual)
Dates: Start 2012-11-09 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2026-01-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (215):
- United States (83):
  - Birmingham, Alabama
  - Gilbert, Arizona
  - Tucson, Arizona
  - Burbank, California
  - Duarte, California
  - Fresno, California
  - Fullerton, California
  - La Jolla, California
  - Long Beach, California
  - Los Angeles, California
  - Sacramento, California
  - San Luis Obispo, California
  - Santa Barbara, California
  - Santa Monica, California
  - Stanford, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Lonetree, Colorado
  - Washington D.C., District of Columbia
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Lawrenceville, Georgia
  - Chicago, Illinois
  - Maywood, Illinois
  - Niles, Illinois
  - Zion, Illinois
  - Fort Wayne, Indiana
  - Goshen, Indiana
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Fairway, Kansas
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Springfield, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Basking Ridge, New Jersey
  - Hackensack, New Jersey
  - Morristown, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Commack, New York
  - New York, New York
  - Rochester, New York
  - Rockville Centre, New York
  - The Bronx, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Bismarck, North Dakota
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Richmond, Virginia
  - Kennewick, Washington
  - Seattle, Washington
  - Vancouver, Washington
  - Yakima, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Australia (11):
  - Kingswood, New South Wales
  - St Leonards, New South Wales
  - Westmead, New South Wales
  - South Brisbane, Queensland
  - Bedford Park, South Australia
  - Hobart, Tasmania
  - East Melbourne, Victoria
  - Geelong, Victoria
  - Heidelberg, Victoria
  - Parkville, Victoria
  - Perth, Western Australia
- Belgium (3):
  - Antwerp
  - Bruges
  - Ghent
- Brazil (6):
  - Salvador, Estado de Bahia
  - Curitiba, Paraná
  - Porto Alegre, Rio Grande do Sul
  - Santo André, São Paulo
  - Rio de Janeiro
  - São Paulo
- Canada (7):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Toronto, Ontario
  - Montreal, Quebec
  - Saskatoon, Saskatchewan
- Czechia (2):
  - Hradec Králové
  - Prague
- Denmark (5):
  - Aalborg
  - Aarhus C
  - Copenhagen
  - Odense C
  - Roskilde
- France (4):
  - Argenteuil, Cedex
  - La Tronche
  - Limoges
  - Paris
- Hong Kong (3):
  - Lai Chi Kok, Kowloon
  - Hong Kong
  - Tuenmen
- Hungary (5):
  - Budapest
  - Debrecen
  - Győr
  - Pécs
  - Szeged
- Italy (13):
  - Modena, Emilia-Romagna
  - Rome, Lazio
  - Alessandria
  - Bologna
  - Cagliari
  - Cuneo
  - Genova
  - Milan
  - Napoli
  - Rionero in Volture
  - Rome
  - Rozzano
  - Torrette Di Ancona
- Japan (10):
  - Higashiku, Fukuoka
  - Minamiku, Fukuoka-city
  - Minamiku, Hiroshima-city
  - Shōwamachi, Maebashi-city
  - Chikusa-ku, Nagoya
  - Suita, Osaka
  - Aoba-ku, Sendai-city
  - Chūōku
  - Isehara-shi
  - Kōtoku
- Norway (2):
  - Bergen
  - Oslo
- Poland (7):
  - Gdansk
  - Katowice
  - Krakow
  - L0dz
  - Olsztyn
  - Warsaw
  - Wroclaw
- Russia (6):
  - Ufa, Bashkortostan Republic
  - Saint Petersburg, Poselok Pesochny
  - Kazan', Republic Tatrstan
  - Moscow
  - Moskva
  - Saint Petersburg
- South Africa (5):
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - eManzimtoti, KwaZulu-Natal
  - Bloemfontein
  - Cape Town
- South Korea (8):
  - Goyang-si, Gyeonggi-do
  - Hwasun-gun, Jeollanam-do
  - Seocho-gu, Seoul
  - Busan
  - Daegu
  - Incheon
  - Jeonju
  - Seoul
- Spain (7):
  - Badalona
  - Barcelona
  - Marbella
  - Pamplona
  - Salamanca
  - Santiago de Compostela
  - Valencia
- Taiwan (5):
  - Changhua
  - Chiayi County 613
  - Tainan
  - Taipei
  - Taoyuan
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Samsun
- United Kingdom (20):
  - Truro, Cornwall
  - Aberdeen, Scotland
  - Glasgow, Scotland
  - Sutton, Surrey
  - Cardiff, Wales
  - Birmingham
  - Canterbury
  - Exeter
  - Inverness
  - Leicester
  - Lincoln
  - Liverpool
  - London
  - Manchester
  - Norfolk
  - Northwood
  - Nottingham
  - Oxford
  - Romford
  - Southampton

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] Crosswell HE, LaCasce AS, Bartlett NL, Straus DJ, Savage KJ, Zinzani PL, Collins GP, Fanale M, Fenton K, Dong C, Miao H, Grigg AP. Brentuximab vedotin with chemotherapy in adolescents and young adults with stage III or IV classical Hodgkin lymphoma in ECHELON-1. Haematologica. 2024 Mar 1;109(3):982-987. doi: 10.3324/haematol.2023.283303. No abstract available. PMID 37794803
- [Derived] Ansell SM, Radford J, Connors JM, Dlugosz-Danecka M, Kim WS, Gallamini A, Ramchandren R, Friedberg JW, Advani R, Hutchings M, Evens AM, Smolewski P, Savage KJ, Bartlett NL, Eom HS, Abramson JS, Dong C, Campana F, Fenton K, Puhlmann M, Straus DJ; ECHELON-1 Study Group. Overall Survival with Brentuximab Vedotin in Stage III or IV Hodgkin's Lymphoma. N Engl J Med. 2022 Jul 28;387(4):310-320. doi: 10.1056/NEJMoa2206125. Epub 2022 Jul 13. PMID 35830649
- [Derived] Evens AM, Connors JM, Younes A, Ansell SM, Kim WS, Radford J, Feldman T, Tuscano J, Savage KJ, Oki Y, Grigg A, Pocock C, Dlugosz-Danecka M, Fenton K, Forero-Torres A, Liu R, Jolin H, Gautam A, Gallamini A. Older patients (aged >/=60 years) with previously untreated advanced-stage classical Hodgkin lymphoma: a detailed analysis from the phase III ECHELON-1 study. Haematologica. 2022 May 1;107(5):1086-1094. doi: 10.3324/haematol.2021.278438. PMID 34162178
- [Derived] Straus DJ, Dlugosz-Danecka M, Connors JM, Alekseev S, Illes A, Picardi M, Lech-Maranda E, Feldman T, Smolewski P, Savage KJ, Bartlett NL, Walewski J, Ramchandren R, Zinzani PL, Hutchings M, Munoz J, Lee HJ, Kim WS, Advani R, Ansell SM, Younes A, Gallamini A, Liu R, Little M, Fenton K, Fanale M, Radford J. Brentuximab vedotin with chemotherapy for stage III or IV classical Hodgkin lymphoma (ECHELON-1): 5-year update of an international, open-label, randomised, phase 3 trial. Lancet Haematol. 2021 Jun;8(6):e410-e421. doi: 10.1016/S2352-3026(21)00102-2. PMID 34048680
- [Derived] Straus DJ, Dlugosz-Danecka M, Alekseev S, Illes A, Picardi M, Lech-Maranda E, Feldman T, Smolewski P, Savage KJ, Bartlett NL, Walewski J, Ramchandren R, Zinzani PL, Hutchings M, Connors JM, Radford J, Munoz J, Kim WS, Advani R, Ansell SM, Younes A, Miao H, Liu R, Fenton K, Forero-Torres A, Gallamini A. Brentuximab vedotin with chemotherapy for stage III/IV classical Hodgkin lymphoma: 3-year update of the ECHELON-1 study. Blood. 2020 Mar 5;135(10):735-742. doi: 10.1182/blood.2019003127. PMID 31945149
- [Derived] Ramchandren R, Advani RH, Ansell SM, Bartlett NL, Chen R, Connors JM, Feldman T, Forero-Torres A, Friedberg JW, Gopal AK, Gordon LI, Kuruvilla J, Savage KJ, Younes A, Engley G, Manley TJ, Fenton K, Straus DJ. Brentuximab Vedotin plus Chemotherapy in North American Subjects with Newly Diagnosed Stage III or IV Hodgkin Lymphoma. Clin Cancer Res. 2019 Mar 15;25(6):1718-1726. doi: 10.1158/1078-0432.CCR-18-2435. Epub 2019 Jan 7. PMID 30617130
- [Derived] Connors JM, Jurczak W, Straus DJ, Ansell SM, Kim WS, Gallamini A, Younes A, Alekseev S, Illes A, Picardi M, Lech-Maranda E, Oki Y, Feldman T, Smolewski P, Savage KJ, Bartlett NL, Walewski J, Chen R, Ramchandren R, Zinzani PL, Cunningham D, Rosta A, Josephson NC, Song E, Sachs J, Liu R, Jolin HA, Huebner D, Radford J; ECHELON-1 Study Group. Brentuximab Vedotin with Chemotherapy for Stage III or IV Hodgkin's Lymphoma. N Engl J Med. 2018 Jan 25;378(4):331-344. doi: 10.1056/NEJMoa1708984. Epub 2017 Dec 10. PMID 29224502
- [Derived] Younes A, Connors JM, Park SI, Fanale M, O'Meara MM, Hunder NN, Huebner D, Ansell SM. Brentuximab vedotin combined with ABVD or AVD for patients with newly diagnosed Hodgkin's lymphoma: a phase 1, open-label, dose-escalation study. Lancet Oncol. 2013 Dec;14(13):1348-56. doi: 10.1016/S1470-2045(13)70501-1. Epub 2013 Nov 15. PMID 24239220

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 218 investigative sites in Asia Pacific, Europe, Latin America, and North America from 09 November 2012 to the primary completion date of 20 April 2017.
Pre-assignment Details: Participants with histologically confirmed diagnosis of advanced classical hodgkin lymphoma (cHL) were enrolled to receive: brentuximab vedotin 1.2 mg/kg plus doxorubicin 25 mg/m^2, vinblastine 6 mg/m^2, and dacarbazine 375 mg/m^2 (A+AVD) or doxorubicin 25 mg/m^2, bleomycin 10 units/m^2, vinblastine 6 mg/m^2, and dacarbazine 375 mg/m^2 (ABVD).
Groups:
- A+AVD: Brentuximab vedotin 1.2 milligram per kilogram (mg/kg), infusion, intravenously over 30-minutes plus doxorubicin 25 milligram per square meter (mg/m^2), vinblastine 6 mg/m^2, and dacarbazine 375 mg/m^2, infusion, intravenously, once on Days 1 and 15 of each 28-day treatment cycle for up to a maximum of 6 cycles. Brentuximab vedotin was administered within approximately 1 hour after completion of AVD.
- ABVD: Doxorubicin 25 mg/m^2, bleomycin 10 units per square meter (units/m^2), vinblastine 6 mg/m^2, and dacarbazine 375 mg/m^2, infusion, intravenously, once on Days 1 and 15 of each 28-day treatment cycle for up to a maximum of 6 cycles.
Period: Overall Study
Arm/Group | A+AVD | ABVD
Started | 664 | 670
Treated | 662 | 659
Completed | 0 | 0
Not Completed | 664 | 670
Not completed — Ongoing | 601 | 586
Not completed — Other | 11 | 11
Not completed — Withdrawal by Subject | 36 | 44
Not completed — Lost to Follow-up | 16 | 29

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants randomized to treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | A+AVD | ABVD | Total
Number analyzed (Participants) | 664 | 670 | 1334
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The ITT population included all participants randomized to treatment.
  years | 38.8 (15.83) | 40.2 (16.05) | 39.5 (15.95)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The ITT population included all participants randomized to treatment.
  Participants
    Female | 286 | 272 | 558
    Male | 378 | 398 | 776
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The ITT population included all participants randomized to treatment.
  Participants
    Hispanic or Latino | 51 | 55 | 106
    Not Hispanic or Latino | 571 | 577 | 1148
    Unknown or Not Reported | 42 | 38 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The ITT population included all participants randomized to treatment.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 56 | 57 | 113
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 20 | 25 | 45
    White | 560 | 554 | 1114
    More than one race | 18 | 17 | 35
    Unknown or Not Reported | 10 | 17 | 27

OUTCOME MEASURES:

1. Primary Outcome: Modified Progression-free Survival (mPFS) Per Independent Review Facility (IRF)
Description: mPFS was defined as the time from the date of randomization to the date of the first of documentation of progressive disease (PD), death due to any cause, or for participants who were confirmed non complete responders per IRF, receipt of subsequent anticancer therapy for Hodgkin lymphoma (HL) after completion of frontline therapy. PD was defined as any new lesion or increase by greater than or equal to (>=) 50 percent (%) of previously involved sites from nadir. Frontline therapy is the part of standard set of treatments.
Time Frame: Baseline until PD or death or receipt of any subsequent anticancer therapy for HL after completion of frontline therapy (approximately up to 4 years)
Population: The ITT population included all participants randomized to treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A+AVD | ABVD
Number analyzed (Participants) | 664 | 670
months | NA [48.2 to NA] — Median and confidence interval was not estimable due to low number of participants with events. | NA [NA to NA] — Median and confidence interval was not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: A+AVD vs ABVD; Hazard ratio (A+AVD/ABVD) and 95% confidence interval (CI) are based on a stratified Cox's proportional hazard regression model with stratification factors region and number of International Prognostic Factor Project (IPFP) risk factors at baseline with treatment as the explanatory variable in the model. Hazard ratio less than (<) 1 favors A+AVD arm; Test type: Superiority; p = 0.035, Log Rank; Hazard Ratio (HR) = 0.770, 95% CI 2-sided [0.603 to 0.983]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death. Participants without documented death at the time of analysis were censored at the date last known to be alive.
Time Frame: Baseline until death (approximately up to 4 years)
Population: The ITT population included all participants randomized to treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A+AVD | ABVD
Number analyzed (Participants) | 664 | 670
months | NA [NA to NA] — Median and confidence interval was not estimable due to low number of participants with events. | NA [NA to NA] — Median and confidence interval was not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: A+AVD vs ABVD; Hazard ratio (A+AVD/ABVD) and 95% CI are based on a stratified Cox's proportional hazard regression model with stratification factors region and number of IPFP risk factors at baseline with treatment as the explanatory variable in the model. Hazard ratio <1 favors A+AVD arm; Test type: Superiority; p = 0.199, Log Rank; Hazard Ratio (HR) = 0.728, 95% CI 2-sided [0.448 to 1.184]

3. Secondary Outcome: Complete Remission (CR) Rate at the End of Randomized Regimen Per IRF
Description: CR rate at the end of randomized regimen per investigator was defined as the percentage of participants who achieved CR at the end of treatment with randomized regimen (ABVD or A+AVD) as determined by IRF. CR was defined as disappearance of all evidence of disease.
Time Frame: Baseline up to end of randomized regimen (approximately 1 year)
Population: The ITT population included all participants randomized to treatment.
Measure: Number; unit: percentage of participants
Arm/Group | A+AVD | ABVD
Number analyzed (Participants) | 664 | 670
percentage of participants | 73 | 70

4. Secondary Outcome: Number of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE) and Serious Adverse Event (SAE)
Time Frame: Baseline up to 30 days after last dose of study drug (approximately 1 year)
Population: The safety population included all enrolled participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | A+AVD | ABVD
Number analyzed (Participants) | 662 | 659
participants
  TEAE | 653 | 646
  SAE | 284 | 178

5. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Values
Time Frame: Baseline up to 30 days after last dose of study drug (approximately 1 year)
Population: The safety population included all enrolled participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | A+AVD | ABVD
Number analyzed (Participants) | 662 | 659
participants | 662 | 658

6. Secondary Outcome: Event-free Survival (EFS) Per IRF
Description: EFS was defined as the time from randomization until any cause of treatment failure: PD, premature discontinuation of randomized treatment for any reason, or death due to any cause, whichever occurs first. PD was defined as any new lesion or increase by >=50% of previously involved sites from nadir per IRF.
Time Frame: Baseline until PD or discontinuation of treatment or death, whichever occurs first (approximately up to 4 years)
Population: The ITT population included all participants randomized to treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A+AVD | ABVD
Number analyzed (Participants) | 664 | 670
months | NA [43.8 to NA] — Median and confidence interval was not estimable due to low number of participants with events. | NA [NA to NA] — Median and confidence interval was not estimable due to low number of participants with events.

7. Secondary Outcome: Disease-free Survival (DFS) Per IRF
Description: DFS per IRF was defined as the time from CR to disease progression as determined by an IRF or to death from lymphoma or acute toxicity from treatment. CR was defined as disappearance of all evidence of disease.
Time Frame: From CR until PD or death (approximately up to 4 years)
Population: The ITT included all participants randomized to treatment. The ITT population where participants achieved CR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A+AVD | ABVD
Number analyzed (Participants) | 543 | 528
months | NA [42.1 to NA] — Median and confidence interval was not estimable due to low number of participants with events. | NA [NA to NA] — Median and confidence interval was not estimable due to low number of participants with events.

8. Secondary Outcome: Overall Response Rate (ORR) Per IRF
Description: ORR per IRF was defined as the percentage of participants who achieved CR or partial remission (PR) at the end of treatment with randomized regimen (ABVD or A+AVD) as determined by an IRF. CR was defined as disappearance of all evidence of disease. PR was defined as regression of measurable disease and no new sites.
Time Frame: Baseline up to end of randomized regimen (approximately 1 year)
Population: The ITT population included all participants randomized to treatment.
Measure: Number; unit: percentage of participants
Arm/Group | A+AVD | ABVD
Number analyzed (Participants) | 664 | 670
percentage of participants | 86 | 83

9. Secondary Outcome: Duration of Response (DOR) Per IRF
Description: DOR per IRF in participants with response was the time between first documentation of response (PR or CR) and PD as determined by an IRF. PD was defined as any new lesion or increase by >=50% of previously involved sites from nadir. CR was defined as disappearance of all evidence of disease. PR was defined as regression of measurable disease and no new sites.
Time Frame: From first documented response until PD (approximately 4 years)
Population: The ITT population included all participants randomized to treatment. The ITT population where participants achieved confirmed response of CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A+AVD | ABVD
Number analyzed (Participants) | 628 | 623
months | NA [42.1 to NA] — Median and confidence interval was not estimable due to low number of participants with events. | NA [NA to NA] — Median and confidence interval was not estimable due to low number of participants with events.

10. Secondary Outcome: Duration of Complete Remission (DOCR) Per IRF
Description: DOCR per IRF in participants with CR was the time between first documentation of CR and PD as determined by an IRF. PD was defined as any new lesion or increase by >=50% of previously involved sites from nadir. CR was defined as disappearance of all evidence of disease.
Time Frame: From first documentation of CR until PD (approximately 4 years)
Population: The ITT population included all participants randomized to treatment. The ITT population where participants achieved CR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A+AVD | ABVD
Number analyzed (Participants) | 543 | 528
months | NA [42.1 to NA] — Median and confidence interval was not estimable due to low number of participants with events. | NA [NA to NA] — Median and confidence interval was not estimable due to low number of participants with events.

11. Secondary Outcome: Percentage of Participants Not in CR Per IRF Who Received Subsequent Radiation After Completion of Frontline Therapy
Description: CR was defined as disappearance of all evidence of disease as determined by an IRF.
Time Frame: Baseline up to end of frontline therapy (approximately 4 years)
Population: The ITT population included all participants randomized to treatment.
Measure: Number; unit: percentage of participants
Arm/Group | A+AVD | ABVD
Number analyzed (Participants) | 664 | 670
percentage of participants | 8 | 13

12. Secondary Outcome: Complete Remission (CR) Per IRF Rate at the End of Frontline Therapy
Description: CR rate at the end of frontline therapy per IRF was defined as the percentage of participants who achieved CR at the end of frontline therapy that is after completion of either randomized regimen or alternate frontline therapy as determined by an IRF. CR was defined as disappearance of all evidence of disease.
Time Frame: Baseline up to end of frontline therapy (approximately 4 years)
Population: The ITT population included all participants randomized to treatment.
Measure: Number; unit: percentage of participants
Arm/Group | A+AVD | ABVD
Number analyzed (Participants) | 664 | 670
percentage of participants | 73 | 71

13. Secondary Outcome: Positron Emission Tomography (PET) Negativity Rate Per IRF at Cycle 2
Description: PET negativity rate at Cycle 2 was defined as the percentage of participants with negative Cycle 2 PET results defined as Deauville score less than or equal to (<=) 3 at Cycle 2. The Deauville score according to IRF assessment of response was used to evaluate the results of PET scans.
Time Frame: Cycle 2 Day 25
Population: The ITT population included all participants randomized to treatment.
Measure: Number; unit: percentage of participants
Arm/Group | A+AVD | ABVD
Number analyzed (Participants) | 664 | 670
percentage of participants | 89 | 86

14. Secondary Outcome: A+AVD: Cmax: Maximum Observed Serum Concentration for Brentuximab Vedotin Antibody-drug Conjugate (ADC) and Total Antibody (TAb)
Time Frame: Cycle 1 Day 1 and Cycle 3 Day 1: pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: The pharmacokinetic (PK) population included enrolled participants with sufficient dosing and PK data to reliably estimate PK parameters as determined by a clinical pharmacologist. The intensive PK (iPK) population was the subset of PK population. The iPK population where data at specified timepoints was available.
Measure: Geometric Mean (Standard Deviation); unit: microgram per milliliter (microgm/mL)
Arm/Group | A+AVD
Number analyzed (Participants) | 59
microgram per milliliter (microgm/mL)
  Cycle 1 Day 1: ADC: number analyzed (Participants) | 55
  Cycle 1 Day 1: ADC | 22.9 (6.72)
  Cycle 3 Day 1: ADC: number analyzed (Participants) | 52
  Cycle 3 Day 1: ADC | 23.6 (6.81)
  Cycle 1 Day 1: TAb: number analyzed (Participants) | 55
  Cycle 1 Day 1: TAb | 22.6 (5.48)
  Cycle 3 Day 1: TAb: number analyzed (Participants) | 52
  Cycle 3 Day 1: TAb | 26.4 (6.11)

15. Secondary Outcome: A+AVD: Cmax: Maximum Observed Plasma Concentration for Brentuximab Vedotin Monomethyl Auristatin E (MMAE)
Time Frame: Cycle 1 Day 1 and Cycle 3 Day 1: pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: The PK population included enrolled participants with sufficient dosing and PK data to reliably estimate PK parameters as determined by a clinical pharmacologist. The iPK population was the subset of PK population. The iPK population where data at specified timepoints was available.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | A+AVD
Number analyzed (Participants) | 59
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 3.20 (2.99)
  Cycle 3 Day 1: number analyzed (Participants) | 56
  Cycle 3 Day 1 | 1.36 (0.790)

16. Secondary Outcome: A+AVD: AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Brentuximab Vedotin ADC and TAb
Time Frame: Cycle 1 Day 1: pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: day*microgram per milliliter (day*ug/mL)
Arm/Group | A+AVD
Number analyzed (Participants) | 59
day*microgram per milliliter (day*ug/mL)
  Cycle 1 Day 1: ADC: number analyzed (Participants) | 53
  Cycle 1 Day 1: ADC | 47.4 (12.0)
  Cycle 1 Day 1: TAb: number analyzed (Participants) | 51
  Cycle 1 Day 1: TAb | 93.0 (25.7)

17. Secondary Outcome: A+AVD: AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Brentuximab Vedotin MMAE
Time Frame: Cycle 1 Day 1: pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: day*nanogram per milliliter (day*ng/mL)
Arm/Group | A+AVD
Number analyzed (Participants) | 59
day*nanogram per milliliter (day*ng/mL) | 25.3 (19.2)

18. Secondary Outcome: A+AVD: Number of Participants With Antitherapeutic Antibody (ATA) and Neutralizing Antitherapeutic Antibody (nATA) Positive for Brentuximab Vedotin
Description: The nATA positive was defined as positive ATA with neutralizing activity at any postbaseline visit.
Time Frame: Baseline up to end of treatment (approximately 1 year)
Population: The safety population included all enrolled participants who received at least 1 dose of any study drug. The safety population-immunogenicity-evaluable participants where baseline and at least one postbaseline sample was available.
Measure: Number; unit: participants
Arm/Group | A+AVD
Number analyzed (Participants) | 632
participants
  ATA positive | 109
  nATA positive | 12

19. Secondary Outcome: Change From Baseline in Patient-Reported Outcome (PRO) Scores by mPFS Based on European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-C30 (EORTC QLQ-C30) at EOT
Description: EORTC QLQ-C30 included 30 items across 5 functional scales (physical, role, cognitive, emotional, and social), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) and global health status/QOL scale. It has 28 questions (4-point scale where 1=not at all [best] to 4=Very Much [worst]) and 2 questions (7-point scale where 1=very poor [worst] to 7= excellent [best]). Raw scores were converted into scale scores from 0 to 100. For functional scales and global health status/QOL scale, higher scores show better QOL; for symptom scales, lower scores show better QOL. mPFS was time from date of randomization to date of first of documentation of PD, death due to any cause, or for participants who were confirmed non complete responders per IRF, receipt of subsequent anticancer therapy for HL after completion of frontline therapy. PD is any new lesion or increase by >=50% of previously involved sites from nadir.
Time Frame: Baseline up to end of treatment (approximately 1 year)
Population: The ITT population included all participants randomized to treatment.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | A+AVD | ABVD
Number analyzed (Participants) | 664 | 670
units on scale
  Baseline: With mPFS event: number analyzed (Participants) | 115 | 143
  Baseline: With mPFS event | 78.15 (16.527) | 76.68 (18.661)
  Without mPFS event: number analyzed (Participants) | 533 | 508
  Without mPFS event | 79.85 (16.648) | 79.91 (16.218)
  Change at end of treatment: with mPFS event: number analyzed (Participants) | 91 | 112
  Change at end of treatment: with mPFS event | 2.68 (15.434) | 8.58 (17.848)
  Change at end of treatment: without mPFS event: number analyzed (Participants) | 475 | 452
  Change at end of treatment: without mPFS event | 3.35 (17.417) | 6.08 (16.141)

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events that started after the first dose of study drug and no more than 30 days (approximately 1 year) for a serious adverse event after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. The safety population included all enrolled participants who received at least 1 dose of any study drug.
Arm/Group | A+AVD | ABVD
All-Cause Mortality (participants affected / at risk) | 9/662 | 13/659
Serious Adverse Events (participants affected / at risk) | 284/662 | 178/659
Other Adverse Events (participants affected / at risk) | 644/662 | 632/659
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A+AVD (N=662) | ABVD (N=659)
Febrile neutropenia (Blood and lymphatic system disorders) | 114 (151) | 43 (52)
Neutropenia (Blood and lymphatic system disorders) | 19 (30) | 4 (5)
Anaemia (Blood and lymphatic system disorders) | 7 (10) | 3 (3)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 18 (19) | 15 (18)
Lung infection (Infections and infestations) | 4 (4) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 14 (15) | 4 (4)
Neutropenic sepsis (Infections and infestations) | 8 (10) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1) | 4 (4)
Septic shock (Infections and infestations) | 4 (6) | 0 (0)
Septic embolus (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 7 (8) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 5 (5) | 2 (2)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 5 (5) | 2 (3)
Pneumocystis jirovecii infection (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 2 (2) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (3) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia viral (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 2 (2) | 0 (0)
Pericoronitis (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 2 (2)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Genital infection female (Infections and infestations) | 0 (0) | 1 (1)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infected lymphocele (Infections and infestations) | 1 (1) | 0 (0)
Phlebitis infective (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Flavivirus infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Moraxella infection (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 44 (55) | 28 (32)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (3)
Pain (General disorders) | 1 (2) | 1 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 2 (2)
Death (General disorders) | 1 (1) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Device related thrombosis (General disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 14 (15) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (11) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (7) | 3 (3)
Constipation (Gastrointestinal disorders) | 11 (12) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 11 (13) | 1 (1)
Colitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 3 (4)
Ileus (Gastrointestinal disorders) | 3 (3) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 4 (5) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 9 (9)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 12 (13)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 10 (10) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 2 (3)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 4 (4)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Brachiocephalic vein occlusion (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (3) | 2 (2)
Lethargy (Nervous system disorders) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (3) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (3) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (3) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 1 (1)
Pseudomonas test positive (Investigations) | 0 (0) | 1 (1)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 2 (2) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Schizoaffective disorder bipolar type (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Branchial cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A+AVD (N=662) | ABVD (N=659)
Neutropenia (Blood and lymphatic system disorders) | 374 (1169) | 291 (813)
Anaemia (Blood and lymphatic system disorders) | 136 (237) | 65 (97)
Leukopenia (Blood and lymphatic system disorders) | 42 (124) | 37 (118)
Nausea (Gastrointestinal disorders) | 346 (673) | 369 (735)
Constipation (Gastrointestinal disorders) | 273 (361) | 239 (336)
Vomiting (Gastrointestinal disorders) | 212 (342) | 183 (284)
Diarrhoea (Gastrointestinal disorders) | 176 (231) | 121 (155)
Stomatitis (Gastrointestinal disorders) | 138 (182) | 104 (135)
Abdominal pain (Gastrointestinal disorders) | 135 (185) | 65 (79)
Dyspepsia (Gastrointestinal disorders) | 84 (100) | 75 (93)
Abdominal pain upper (Gastrointestinal disorders) | 64 (74) | 34 (37)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 33 (36) | 47 (49)
Fatigue (General disorders) | 209 (272) | 211 (293)
Pyrexia (General disorders) | 149 (224) | 128 (191)
Asthenia (General disorders) | 65 (97) | 42 (66)
Chills (General disorders) | 37 (52) | 46 (51)
Non-cardiac chest pain (General disorders) | 37 (40) | 45 (53)
Upper respiratory tract infection (Infections and infestations) | 68 (76) | 69 (75)
Nasopharyngitis (Infections and infestations) | 28 (39) | 35 (40)
Weight decreased (Investigations) | 148 (168) | 40 (46)
Neutrophil count decreased (Investigations) | 86 (285) | 78 (191)
Alanine aminotransferase increased (Investigations) | 68 (92) | 26 (28)
White blood cell count decreased (Investigations) | 46 (81) | 34 (59)
Aspartate aminotransferase increased (Investigations) | 47 (58) | 19 (21)
Gamma-glutamyltransferase increased (Investigations) | 34 (41) | 10 (13)
Decreased appetite (Metabolism and nutrition disorders) | 118 (156) | 76 (106)
Hypokalaemia (Metabolism and nutrition disorders) | 45 (50) | 24 (35)
Hyperglycaemia (Metabolism and nutrition disorders) | 34 (44) | 14 (18)
Bone pain (Musculoskeletal and connective tissue disorders) | 125 (200) | 66 (87)
Arthralgia (Musculoskeletal and connective tissue disorders) | 89 (113) | 77 (98)
Myalgia (Musculoskeletal and connective tissue disorders) | 80 (127) | 70 (87)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 79 (108) | 67 (93)
Back pain (Musculoskeletal and connective tissue disorders) | 82 (96) | 49 (59)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 40 (48) | 29 (34)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 36 (41) | 17 (18)
Peripheral sensory neuropathy (Nervous system disorders) | 189 (298) | 111 (149)
Neuropathy peripheral (Nervous system disorders) | 174 (261) | 85 (103)
Headache (Nervous system disorders) | 93 (124) | 92 (117)
Paraesthesia (Nervous system disorders) | 84 (120) | 73 (89)
Dizziness (Nervous system disorders) | 64 (74) | 57 (65)
Dysgeusia (Nervous system disorders) | 48 (52) | 48 (68)
Peripheral motor neuropathy (Nervous system disorders) | 40 (50) | 8 (9)
Insomnia (Psychiatric disorders) | 126 (134) | 82 (89)
Anxiety (Psychiatric disorders) | 50 (53) | 49 (52)
Depression (Psychiatric disorders) | 35 (36) | 25 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 97 (108) | 122 (139)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 79 (97) | 121 (136)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 72 (82) | 55 (65)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 40 (41) | 28 (31)
Alopecia (Skin and subcutaneous tissue disorders) | 173 (194) | 146 (165)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 43 (60) | 28 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2015-03-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT01712490/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT01712490/SAP_001.pdf